CLINICAL TRIAL: NCT01286610
Title: Application of Vibration Therapy as a Measure of Muscle Activation in ICU Patients and Its Effect on Hemodynamics, Intracranial Pressure as Well as Energy Metabolism
Brief Title: Applicability and Safety of Vibration Therapy in Intensive Care Unit (ICU) Patients
Acronym: VTICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Steffen Weber-Carstens, Dr. med. Steffen Weber-Carstens, Dept. of Anesthesiology and Intensive Care Medicine, Charite University, Berlin, Germany., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KFO192/2-P3-Vibro-01
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Respiratory Failure; Sepsis; Brain Injury
Keywords: vibration; ICU; blood pressure; intracranial pressure; infection; indirect calorimetry
MeSH Terms: conditions — Respiratory Insufficiency; Sepsis; Brain Injuries; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vibration therapy and electrical muscle stimulation (Other)
  Interventions: Device: ProMedVi Vibrosphere; Device: schwa-medico MUSKELaktiv; Device: Galileo Home Plus (ICU)

INTERVENTIONS:
Device: ProMedVi Vibrosphere — vibration therapy
Device: schwa-medico MUSKELaktiv — Electrical muscle stimulation
Device: Galileo Home Plus (ICU) — vibration therapy

SUMMARY:
Vibration therapy is used for different indications in rehabilitation and sports medicine. So far, vibration therapy has not been investigated within the ICU setting. The investigators created this setting to show safety and applicability of vibration therapy in ICU patients. 30 patients will be stimulated by vibration therapy on two separate days during their ICU stay. Three collectives of equal size will be observed: One with patients on mechanical ventilation without signs of infection or suspected intracranial pressure problems, a second one with patients on mechanical ventilation in addition to signs of systemic inflammation but absence of suspected intracranial pressure problems, and a third one with patients on mechanical ventilation, signs of systemic inflammation in addition to presence of controlled intracranial pressure problems. Typical parameters of hemodynamic status, intracranial pressure and energy metabolism will be recorded for a defined period of time before, during and after vibration therapy itself. Vibration therapy will be combined with protocol based physiotherapy.

Our aim is to show the effects of vibration therapy in ICU patients and its safe applicability.

ADDITION 06th of May 2011: Additionally we will perform euglycaemic hyperinsulinemic clamp and intervention on one day of ICU stay in 20 patients. Under clamp conditions we will perform a vibration therapy (ProMedVi Vibrosphere™) on patients' legs. On top we will perform electrical muscle stimulation (schwa-medico, MUSKELaktiv™) on one ventral upper leg, randomized chosen. Measuring the local skeletal muscle metabolism will be done by microdialysis in Vastus lateralis on both sides - comparing vibration therapy and vibration therapy combined with electrical muscle stimulation.

ELIGIBILITY:
Inclusion Criteria:

* immobilized icu patients:

  * with mechanical ventilation without signs of infection
  * with mechanical ventilation and SIRS or sepsis
  * with mechanical ventilation, with controlled elevated intracranial pressure and with or without SIRS or sepsis
* signed declaration of consent by the patient or its legal proxy

Exclusion Criteria:

* age < 18 years old
* already known neuromuscular disease
* missing declaration of consent by the patient or its legal proxy
* implanted heart pacemaker or defibrillator
* pregnancy
* acute thrombosis
* not yet healed fracture ad the part of the body which will be trained
* implants ad the part of the body which will be trained
* a nearly done ophthalmic surgery
* acute disc prolapse
* infaust prognosis, that means death is expected into the next couple of hours, although maximum therapy is done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change of vital parameters as a measure of hemodynamic stability to show safety and tolerability | Continuous record for 90 minutes - within 4 blood samples - vibration therapy compared to baseline
  Changes in heart rate, arterial blood pressure, saturation of peripheral pulse oximetry, intracranial pressure, mechanical ventilation parameters, electrolytes, blood sugar and lactate levels, blood pH, PICCO-parameters, body temperature as well as pO2 und pCO2 partial pressure.

SECONDARY OUTCOMES:
Change of vital parameters as a measure of hemodynamic stability to show safety and tolerability. | Continuous record for 90 minutes - within 4 blood samples - vibration therapy compared to baseline
  Change in heart rate, arterial blood pressure, saturation of peripheral pulse oximetry, intracranial pressure, mechanical ventilation parameters, electrolyte, blood sugar and lactate levels, blood pH, PICCO-parameters, body temperature as well as pO2 und pCO2 partial pressure.
Change in peripheral energy metabolism and hormonal state as a measure of muscle activation and systemic inflammatory reaction induced by vibration therapy. | Continuous record for 90 minutes - within 4 blood samples - vibration therapy compared to baseline
  Change in Parameters of indirect calorimetry, circulating IGF-1, IGFBP-1, IGFBP-3, IL-6, IL-10, insulin, cortisol, blood sugar and lactate levels, blood pH, PICCO-parameters, body temperature as well as pO2 und pCO2 partial pressure.
Change in peripheral energy metabolism and hormonal state as measure of muscle activation and systemic inflammatory reaction induced by vibration therapy | Continuous record for 90 minutes - within 4 blood samples - vibration therapy compared to baseline
  Change in Parameters of indirect calorimetry, circulating IGF-1, IGFBP-1, IGFBP-3, IL-6, IL-10, insulin, cortisol, blood sugar and lactate levels, blood pH, PICCO-parameters, body temperature as well as pO2 und pCO2 partial pressure
Change in systemic and local energy metabolism as measure of muscle activation by vibration therapy and electrical muscle stimulation | Continuous record for app. 10 hours - therapy compared to baseline
  Change in Parameters of indirect calorimetry, circulating IGF-1, IGFBP-1, IGFBP-3, IL-6, IL-10, insulin, cortisol, blood sugar and lactate levels, blood pH, PICCO-parameters, body temperature as well as pO2 und pCO2 partial pressure for systemic energy metabolism. For local skeletal muscle metabolism we will measure glucose, lactate, pyruvate, urea and glycerol by microdialyses technic.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Weber-Carstens, MD, Principal Investigator — Dept. of Anesthesiology and Intensive Care Medicine, Charite University, Berlin, Germany
Locations (1):
- Charite University, Berlin, Germany, Berlin, Germany

REFERENCES:
- [Result] Wollersheim T, Haas K, Wolf S, Mai K, Spies C, Steinhagen-Thiessen E, Wernecke KD, Spranger J, Weber-Carstens S. Whole-body vibration to prevent intensive care unit-acquired weakness: safety, feasibility, and metabolic response. Crit Care. 2017 Jan 9;21(1):9. doi: 10.1186/s13054-016-1576-y. PMID 28065165